CLINICAL TRIAL: NCT01187498
Title: Behavioral Treatment of Overactive Bladder in Men
Acronym: MOTIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B3083-R
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-12

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Behavioral treatment; Drug therapy; Lower urinary tract symptoms; Urinary incontinence; Clinical trial
MeSH Terms: conditions — Urinary Bladder, Overactive; Lower Urinary Tract Symptoms; Urinary Incontinence | interventions — Behavior Therapy; oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Training (Experimental): Behavioral training using delayed voiding, urge suppression techniques, and pelvic floor muscle training
  Interventions: Behavioral: Behavioral training
- Drug Therapy (Active Comparator): Oxybutynin chloride, extended-release, individually-titrated, 5-30 mg
  Interventions: Drug: Oxybutynin chloride, extended-release

INTERVENTIONS:
Behavioral: Behavioral training — Comprehensive behavioral training program using delayed voiding, urge suppression techniques, pelvic floor muscle training, and monitoring with bladder diaries. Treatment is implemented by a nurse practitioner in 4 clinic visits over 8 weeks.
  Other Names: Behavioral treatment
  Arms: Behavioral Training
Drug: Oxybutynin chloride, extended-release — Individually titrated, extended-release oxybutynin chloride, initiated at 10 mg, fluid management handout, and monitoring with bladder diaries. Treatment is implemented by a nurse practitioner in 4 clinic visits over 8 weeks.
  Other Names: Antimuscarinic medication
  Arms: Drug Therapy

SUMMARY:
The primary purpose of this project is to evaluate the effectiveness of behavioral treatment compared to standard drug therapy for symptoms of OAB in male veterans.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a very common and bothersome condition manifested by urgency, frequent urination, urge urinary incontinence, and nocturia. Drug therapy with oxybutynin or tolterodine is the most common approach to treatment of OAB in VA Medical Center clinics and is the standard of care nationally. Although it improves symptoms of OAB for many patients, drug therapy often has side effects, which cause a significant number of patients to discontinue therapy. Further, many symptoms are not completely controlled, even while patients are on the medication. Therefore, there is a need to improve interventions for this common problem. Although behavioral treatment is a well-established treatment for urge urinary incontinence and frequency in women, there are no controlled trials of behavioral treatment for symptoms of OAB in men. The primary purpose of this project is to evaluate the effectiveness of behavioral treatment for symptoms of OAB in male veterans.

The study is a two-site (Birmingham and Atlanta) randomized clinical trial to evaluate the effects of behavioral training compared to a standard (drug) treatment control condition. Subjects are 143 men with OAB as manifested by urgency and frequent urination (>8 voids per day), with or without incontinence, and without significant bladder outlet obstruction. Following a run-in period in which all patients are treated with an alpha blocker to empirically treat any undetected obstruction, they are stratified on severity and presence of urge incontinence and randomized to 8 weeks of behavioral treatment or drug therapy. The behavioral treatment is a comprehensive, behavioral training program, which includes pelvic floor muscle rehabilitation, self monitoring with bladder diaries, and teaching urge suppression and other skills to inhibit detrusor contraction, thus reducing urgency, frequency, incontinence, and nocturia. Patients in the control group receive standard therapy consisting of individually titrated, extended-release oxybutynin, a well-established pharmacologic agent with a state of the art drug delivery system that has the lowest rates of side effects. Bladder diaries completed by subjects prior to randomization and following the last treatment session are used to calculate changes in frequency of urination, as well as other symptoms of overactive bladder, including reports of urgency, incontinence, and nocturia. Secondary outcome measures include patient global ratings of satisfaction and improvement, impact of incontinence, and the American Urological Association (AUA) Symptom Index.

The second purpose of the study is to examine combined behavioral and drug therapy. Following post-treatment assessment, patients who do not achieve satisfactory outcomes with either behavioral or drug therapy alone are crossed over into a second phase, in which they receive combined treatment to improve outcome as much as possible.

This study will yield important information related to alternative treatment of OAB in male veterans. Though many clinicians use drug therapy routinely in the treatment of OAB, most do not offer behavioral treatments such as pelvic floor muscle training for this problem. Thus, this study has potential to alter standards of care for OAB in men.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Community-dwelling
* Veteran
* Self-reported urgency
* Self-reported frequent urination
* Mean of > 8 voids per 24-hour day on bladder diary
* Able to come to clinic

Exclusion Criteria:

* Urologic surgery in the past 6 months
* Nonambulatory (unless has independent transfer skills)
* Flow rate < 5mL at baseline and < 10mL/sec after run-in (on simple uroflowmetry)
* Post-void residual urine volume > 250mL at baseline and > 150mL after run-in (on bladder ultrasound)
* Continual leakage
* Urinary tract infection (growth of > 100,000 colonies per ml of a urinary pathogen on urine culture). May be reconsidered after treatment and negative culture.
* Fecal impaction
* Poorly controlled diabetes (glycosylated hemoglobin >9 within last 3 months)
* Hematuria on microscopic examination in the absence of infection
* Any unstable medical condition (particularly: decompensated congestive heart failure, malignant arrhythmias, unstable angina)

  -- Impaired mental status (< 24 on Folstein's Mini-Mental State Exam)
* Narrow angle glaucoma
* Gastric retention (by medical history)
* Hypersensitivity to tamsulosin or oxybutynin
* Current use of anticholinergic agents for detrusor instability. May be reconsidered after 2-week wash-out.
* If on diuretic, dose has not been stable for at least three months
* Sleep apnea, unless surgically corrected

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2005-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L. Burgio, PhD MA BA, Principal Investigator — Birmingham, Alabama VA Medical Center
Locations (2):
- United States (2):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia

REFERENCES:
- [Result] Burgio KL, Goode PS, Johnson TM, Hammontree L, Ouslander JG, Markland AD, Colli J, Vaughan CP, Redden DT. Behavioral versus drug treatment for overactive bladder in men: the Male Overactive Bladder Treatment in Veterans (MOTIVE) Trial. J Am Geriatr Soc. 2011 Dec;59(12):2209-16. doi: 10.1111/j.1532-5415.2011.03724.x. Epub 2011 Nov 7. PMID 22092152
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598
- [Derived] Johnson TM 2nd, Markland AD, Goode PS, Vaughan CP, Colli JL, Ouslander JG, Redden DT, McGwin G, Burgio KL. Efficacy of adding behavioural treatment or antimuscarinic drug therapy to alpha-blocker therapy in men with nocturia. BJU Int. 2013 Jul;112(1):100-8. doi: 10.1111/j.1464-410X.2012.11736.x. Epub 2013 Feb 28. PMID 23448285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through mailed surveys about bladder symptoms and through clinics at two Veterans Affairs Medical Centers(2005-2009).
Pre-assignment Details: To minimize possible effect of undetected obstruction we used a 4-week alpha-blocker run-in (tamsulosin 0.4 mg/d or alternative). Participants who continued to meet inclusion criteria after run-in were randomized. Alpha-blocker therapy was continued throughout the trial, unless not tolerated.
Groups:
- Behavioral Training: Delayed voiding, urge suppression techniques, pelvic floor muscle training
- Drug Therapy: Individually titrated, extended-release oxybutynin chloride, 5-30mg
Period: Overall Study
Arm/Group | Behavioral Training | Drug Therapy
Started | 73 | 70
Completed | 64 | 60
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Drug Therapy: Individually titrated, extended release oxybutynin chloride
- Total: Total of all reporting groups
Arm/Group | Behavioral Training | Drug Therapy | Total
Number analyzed (Participants) | 73 | 70 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.3) | 64.8 (9.6) | 64.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 73 | 70 | 143
Region of Enrollment [Number; unit: participants]
  United States | 73 | 70 | 143

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Voiding Frequency
Description: Mean voiding frequency per 24 hours derived from 7-day bladder dairy
Time Frame: post-treatment (week 8)
Population: Treatment completers
Measure: Mean (Standard Deviation); unit: voids per 24-hour day
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 64 | 60
voids per 24-hour day | 9.1 (2.5) | 9.5 (2.4)
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; The primary analysis was an equivalence analysis to compare the two treatment groups on posttreatment 24- hour voiding frequency using a margin of ±15% of the drug group mean. Schuirmann's two one-sided tests (TOST) approach was used first to examine completers and then repeated using last observation carried forward to include participants who did not complete therapy. Adjusting the test to regression, the analyses were repeated using baseline voiding frequency as a covariate; Test type: Non-Inferiority or Equivalence — A power analysis indicated that a sample size of 70 per group would provide 80% power with a one-sided alpha of 0.05 to declare two means equivalent, assuming a mean voiding frequency of 8.2 for behavioral treatment, a mean voiding frequency of 8.0 for drug therapy, and a standard deviation of 2.3 for both groups. Equivalence was defined as ±15% of the drug therapy posttreatment mean; p = .001, Regression, Linear; Difference of the Means = .4, Standard Error of Mean 0.346 — The estimated parameter of dispersion is the standard error of the regression coefficient which measured the adjusted difference of the group means

2. Secondary Outcome: Change in Nocturia Frequency
Description: Change in frequency of nocturia episodes based on 7-day bladder diary
Time Frame: baseline to post-treatment (week 8)
Measure: Mean (Standard Deviation); unit: nocturia episodes per night
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 64 | 60
nocturia episodes per night | -0.70 (.72) | -.32 (1.28)
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Standard regression methods adjusting for baseline values; Test type: Superiority or Other; p = .05, Regression, Linear; Difference of the Means = -.38, Standard Error of Mean .188 — The estimated parameter of dispersion represents the standard error for the difference of the group means

3. Secondary Outcome: Change in Urgency Severity
Description: Indevus Urgency Severity Scale incorporated into the 7-day bladder diary. Scores for urgency severity ranged from 0 to 3:
  0: None-no urgency
  1. Mild-awareness of urgency, but is easily tolerated.
  2. Moderate-enough urgency discomfort that it interferes with or shortens usual activity
  3. Severe-extreme urgency discomfort that abruptly stops all activities or tasks.
Time Frame: baseline to post-treatment (week 8)
Population: Participants who completed treatment and returned bladder diary with useable urgency scores
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 61 | 60
Score on scale | .04 (.58) | -.15 (.42)
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Standard regression methods adjusting for baseline values; Test type: Superiority or Other; p = .05, t-test, 2 sided; Difference of Group Means = 0.19, Standard Error of Mean .091 — The estimated parameter of dispersion represents the standard error for the difference of the group means

4. Secondary Outcome: Percent Change in Frequency of Urge Incontinence
Description: Percent change in frequency of urge incontinence episodes based on 7-day bladder diary. Percent change was calculated as ([frequency at baseline] - [frequency at 8 weeks]) / (frequency at baseline).
Time Frame: baseline to post-treatment (week 8)
Population: Included participants who experienced incontinence at baseline only
Measure: Mean (Standard Deviation); unit: Percent change in episodes per week
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 22 | 24
Percent change in episodes per week | 87.2 (.25) | 75.6 (.36)
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Standard regression methods adjusting for baseline values; Test type: Superiority or Other; p = .33, t-test, 2 sided; Difference in Group Means = -.14, Standard Error of Mean 0.091 — The estimated parameter of dispersion represents the standard error for the difference of the group means

5. Secondary Outcome: Change on American Urological Association (AUA) Symptom Index
Description: Change in score on American Urological Association (AUA) Symptom Index (baseline to week 8). The index measures lower urinary tract symptoms. Scores range from 0 to 35, with higher scores indicating worse symptoms.
Time Frame: baseline to post-treatment (week 8)
Population: Completers
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 64 | 60
Scores on the scale | 3.4 (4.6) | 3.2 (5.6)
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Standard regression methods adjusting for baseline values; Test type: Superiority or Other; p = .84, t-test, 2 sided; Median Difference (Net) = 0.20, Standard Error of Mean 0.924 — The estimated parameter of dispersion represents the standard error for the difference of the group means

6. Secondary Outcome: Patient Global Perception of Improvement (GPI)
Description: Patient global perception of improvement ("much better" to "much worse")
Time Frame: post-treatment (week 8)
Population: Completers minus one missing value
Measure: Number; unit: participants
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 63 | 60
participants
  Much better | 23 | 18
  Better | 30 | 34
  About the same | 10 | 7
  Worse | 0 | 1
  Much worse | 0 | 0
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Cochran Mantel-Haenszel procedure used to account for the ordinal nature of responses; Test type: Superiority or Other; p = .69, Cochran-Mantel-Haenszel; Difference in Weighted Group Means = -.0563, Standard Error of Mean .1249 — The estimated parameter of dispersion represents the standard error for the difference of the weighted group means

7. Secondary Outcome: Patient Satisfaction
Description: Patient global rating of satisfaction with progress in treatment ("completely satisfied" to "very dissatisfied")
Time Frame: post-treatment (week 8)
Population: Completers minus one missing value
Measure: Number; unit: participants
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 63 | 60
participants
  Completely satisfied | 36 | 25
  Somewhat satisfied | 25 | 33
  Somewhat dissatisfied | 2 | 2
  Very Dissatisfied | 0 | 0
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Cochran Mantel-Haenszel procedure used to account for the ordinal nature of responses; Test type: Superiority or Other; p = .16, Cochran-Mantel-Haenszel; Difference between Group Weighted Means = -.1563, Standard Error of Mean 0.1009 — The estimated parameter of dispersion represents the standard error for the difference of the weighted group means

8. Secondary Outcome: Patient Global Rating of Activity Restriction
Description: Patient global rating of activity restriction ("not at all" to "all the time")
Time Frame: post-treatment (week 8)
Population: Com0leters minus one missing value
Measure: Number; unit: participants
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 63 | 60
participants
  Not at all | 29 | 31
  Slightly | 19 | 15
  Some of the time | 11 | 13
  All the time | 4 | 1
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Cochran Mantel-Haenszel procedure used to account for the ordinal nature of responses; Test type: Superiority or Other; p = .56, Cochran-Mantel-Haenszel; Difference in Weighted Group Means = 0.1079, Standard Error of Mean .1625 — The estimated parameter of dispersion represents the standard error for the difference of the weighted group means

9. Secondary Outcome: Patient Report of Symptom Distress
Description: Patient report of how disturbed they were by symptoms ("not at all" to "extremely")
Time Frame: post-treatment (week 8)
Population: Completers minos one missing value
Measure: Number; unit: participants
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 63 | 60
participants
  Not at all | 19 | 17
  Slightly | 30 | 35
  Somewhat | 14 | 7
  All the time | 0 | 1
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Cochran Mantel-Haenszel procedure used to account for the ordinal nature of responses; Test type: Superiority or Other; p = .65, Cochran-Mantel-Haenszel; Difference in Weighted Group Means = 0.0540, Standard Error of Mean .1265 — The estimated parameter of dispersion represents the standard error for the difference of the weighted group means

10. Secondary Outcome: Patient Global Rating of Bothersomeness of Side Effects
Description: Patient global rating of how bothersome their side effects were ("no side effects" to "extremely bothersome")
Time Frame: post-treatment (week 8)
Population: Completers minus one missing value
Measure: Number; unit: participants
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 63 | 60
participants
  No side effects | 23 | 11
  Not at all bothersome | 16 | 13
  A Little | 16 | 19
  Somewhat | 7 | 13
  Extremely | 1 | 4
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Cochran Mantel-Haenszel procedure used to account for the ordinal nature of responses; Test type: Superiority or Other; p = .01, Cochran-Mantel-Haenszel

11. Secondary Outcome: Patient Desire for Alternate Treatment
Description: Patient response to "Do you wish to receive another form of treatment?" (yes)
Time Frame: post-treatment (week 8)
Population: Completers minus one missing value
Measure: Number; unit: participants
Arm/Group | Behavioral Training | Drug Therapy
Number analyzed (Participants) | 63 | 60
participants | 18 | 30
Statistical Analysis 1: Comparison: Behavioral Training vs Drug Therapy; Cochran Mantel-Haenszel procedure; Test type: Superiority or Other; p = .02, Chi-squared; Difference in Group Proportions = -.21, Standard Error of Mean .086 — The estimated parameter of dispersion represents the standard error for the difference of the group proportions

ADVERSE EVENTS:
Time Frame: 8-week treatment period
Arm/Group | Behavioral Training | Drug Therapy
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/70
Other Adverse Events (participants affected / at risk) | 0/73 | 0/70

LIMITATIONS AND CAVEATS:
Results can only be generalized to men without evidence of obstruction as determined by uroflowmetry, post-void residual urine (PVR) volume, and a trial of an alpha-blocker.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No